CLINICAL TRIAL: NCT01364207
Title: The Effects of Caffeinated Coffee on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 09-06-052
Record Dates: First submitted 2010-11-05; First posted 2011-06-02 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeinated Coffee 1st Visit, Decaffeinated Coffee 2nd Visit (Experimental): Participants will be given an 8 oz cup of caffeinated coffee on their first visit and 8 oz cup of decaffeinated coffee on their second visit.
  Interventions: Other: Caffeinated Coffee; Other: Decaffeinated Coffee
- Decaffeinated Coffee 1st Visit, Caffeinated Coffee 2nd Visit (Experimental): Participants will be given an 8 oz cup of decaffeinated coffee on their first visit and 8 oz cup of caffeinated coffee on their second visit.
  Interventions: Other: Caffeinated Coffee; Other: Decaffeinated Coffee

INTERVENTIONS:
Other: Caffeinated Coffee — Participants will drink one 8 oz cup in the morning hours. Participants have 15 minutes to drink the coffee but may do so in less time.
Other: Decaffeinated Coffee — Participants will drink one 8 oz cup in the morning hours. Participants have 15 minutes to drink the coffee but may do so in less time.

SUMMARY:
High intraocular pressure (IOP) is a known risk factor for developing primary open-angle glaucoma (POAG). There is controversy in the literature regarding the degree to which caffeine influences IOP, with some studies reporting minimal changes in IOP while others report up to 4 mmHg increases. To date there are no double-masked randomized controlled trials that examine acute caffeinated coffee's effects on IOP in patients with or at risk for primary open-angle glaucoma. The investigators aim to better understand the relationship between acute caffeinated coffee (vs decaffeinate coffee) consumption and IOP in a double-masked, crossover randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 40-89 yrs
* POAG for cases or no forms of glaucoma for controls
* Willingness to drink coffee
* Consent signed

Exclusion Criteria:

* Age less than 40 or greater than 89 yrs
* all forms of glaucoma other than POAG
* any condition inappropriate for tonometry (ie corneal disease, LASIK)
* unable or unwilling to give consent
* unable or unwilling to drink coffee
* pregnancy

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis R Pasquale, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caffeinated Coffee 1st Visit, Decaffeinated Coffee 2nd Visit: Participants drank an 8 oz cup of caffeinated coffee on the their first visit, and then an 8 oz cup of decaffeinated coffee on their second visit. The second visit was completed 2 days to 4 weeks after the first visit, depending on the participants' schedules. Participants did not ingest caffeine in any form starting from 12:01am the day of the visit until after the visit that day except for the study coffee we gave to them.
- Decaffeinated Coffee 1st Visit, Caffeinated Coffee 2nd Visit: Participants drank an 8 oz cup of decaffeinated coffee on the their first visit, and then an 8 oz cup of caffeinated coffee on their second visit. The second visit was completed 2 days to 4 weeks after the first visit, depending on the participants' schedules. Participants did not ingest caffeine in any form starting from 12:01am the day of the visit until after the visit that day except for the study coffee we gave to them.
Period: First Visit (~1.5-2 Hours)
Arm/Group | Caffeinated Coffee 1st Visit, Decaffeinated Coffee 2nd Visit | Decaffeinated Coffee 1st Visit, Caffeinated Coffee 2nd Visit
Started | 54 | 58
Completed | 54 | 58
Not Completed | 0 | 0
Period: Time Between Visits (2 Days to 4 Weeks)
Arm/Group | Caffeinated Coffee 1st Visit, Decaffeinated Coffee 2nd Visit | Decaffeinated Coffee 1st Visit, Caffeinated Coffee 2nd Visit
Started | 54 | 58
Completed | 52 | 54
Not Completed | 2 | 4
Period: Second Visit (~1.5-2 Hours)
Arm/Group | Caffeinated Coffee 1st Visit, Decaffeinated Coffee 2nd Visit | Decaffeinated Coffee 1st Visit, Caffeinated Coffee 2nd Visit
Started | 52 | 54
Completed | 52 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Who Completed Both Study Visits: Only those 106 participants who completed both study visits were included in baseline and final data analyses. The 6 participants who did not complete both study visits were not included in any baseline or final data analyses.
Arm/Group | All Participants Who Completed Both Study Visits
Number analyzed (Participants) | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 52
Baseline Intraocular Pressure on Caffeinated Coffee Visit [Mean (Standard Deviation); unit: mmHg] — The intraocular pressure measured at baseline prior to ingestion of caffeinated coffee on the caffeinated coffee visit.
  mmHg | 15.90 (2.78)
Baseline Intraocular Pressure on Decaffeinated Coffee Visit [Mean (Standard Deviation); unit: mmHg] — The intraocular pressure measured at baseline prior to ingestion of decaffeinated coffee on the decaffeinated coffee visit.
  mmHg | 16.01 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure at 60 Minutes
Description: At the caffeinated coffee visit: Change in intraocular pressure at 60 minutes = intraocular pressure at 60 minutes post caffeinated coffee ingestion minus intraocular pressure at baseline prior to caffeinated coffee ingestion
  At the decaffeinated coffee visit: Change in intraocular pressure at 60 minutes = intraocular pressure at 60 minutes post decaffeinated coffee ingestion minus intraocular pressure at baseline prior to decaffeinated coffee ingestion
Time Frame: Prior to coffee ingestion (baseline), 60 minutes post coffee ingestion
Population: Only those 106 participants who completed both study visits were included in baseline and final data analyses. The 6 participants who did not complete both study visits were not included in any baseline or final data analyses.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Caffeinated Coffee: Participants drank an 8 oz cup of caffeinated coffee.
- Decaffeinated Coffee: Participants drank an 8 oz cup of decaffeinated coffee.
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee
Number analyzed (Participants) | 106 | 106
mm Hg | 1.51 (1.54) | 0.52 (1.29)

2. Primary Outcome: Change in Intraocular Pressure at 90 Minutes
Description: At the caffeinated coffee visit: Change in intraocular pressure at 90 minutes = intraocular pressure at 90 minutes post caffeinated coffee ingestion minus intraocular pressure at baseline prior to caffeinated coffee ingestion
  At the decaffeinated coffee visit: Change in intraocular pressure at 90 minutes = intraocular pressure at 90 minutes post decaffeinated coffee ingestion minus intraocular pressure at baseline prior to decaffeinated coffee ingestion
Time Frame: Prior to coffee ingestion (baseline), 90 minutes post coffee ingestion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee
Number analyzed (Participants) | 106 | 106
mm Hg | 1.46 (1.68) | 0.40 (1.37)

ADVERSE EVENTS:
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/110
Other Adverse Events (participants affected / at risk) | 0/108 | 0/110

LIMITATIONS AND CAVEATS:
We gave subjects caffeinated coffee on one visit and decaffeinated coffee on the other visit. The changes in outcome parameters we observed (ie IOP changes) could be due to other non-caffeine components in the coffee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes